CLINICAL TRIAL: NCT07299864
Title: Non-Operative Management in Patients With Iatrogenic Colorectal Perforations: A Retrospective Multicenter Study
Brief Title: Non-Operative Management in Patients With Iatrogenic Colorectal Perforations
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Taras V. Nechay, Professor of Surgery, Pirogov Russian National Research Medical University
Other Study IDs: 3
Record Dates: First submitted 2025-12-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Iatrogenic Colorectal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the nonoperative management group
- the surgical treatment group

SUMMARY:
This is a retrospective, multicenter observational study that aims to evaluate the efficacy and safety of non-operative management in patients with iatrogenic colorectal perforations.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 years or older

  * Iatrogenic colorectal perforation confirmed during or after diagnostic or therapeutic colonoscopy.

Exclusion Criteria:

* • Patients diagnosed with colorectal perforations due to trauma, acute diverticulitis, anastomotic dehiscence or surgical interventions not related to diagnostic or therapeutic colonoscopy

  * Incomplete records or missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed iatrogenic colorectal perforations occurring during diagnostic or therapeutic colonoscopy at three high-volume tertiary care hospitals
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
survival rate | up to 30 days

SECONDARY OUTCOMES:
occurrence of complications classified according to the Clavien-Dindo | up to 30 days
length of hospital stay | up to 30 days
need for ICU admission | up to 30 days
duration of ICU stay | up to 30 days
stoma formation rate | up to 30 days
re-operation rate | up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov 1 City Clinical Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided